CLINICAL TRIAL: NCT06611319
Title: ENhanced Recovery and ABbreviated LEngth of Anticoagulation for Thromboprophylaxis After Primary Hip Arthroplasty
Acronym: ENABLE-Hip
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prof. Stavros Konstantinides, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Stavros Konstantinides, MD, Univ.-Prof., Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23-01496; 2023-507490-18-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Hip Arthroplasty, Total; Prevention of Venous Thromboembolism
Keywords: Thromboprophylaxis after hip surgery; Rivaroxaban; Abbreviated length of Anticoagulation; Enhanced recovery after surgery; Fast-track surgery; Early mobilization; Pulmonary embolism; Deep vein thrombosis
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis | interventions — Rivaroxaban; N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Intervention Model Description: Investigator-initiated and academically sponsored multicenter randomized double blind active-control non-inferiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abbreviated lenght of thromboprophylaxis (Experimental): Rivaroxaban from day 3-10; Placebo from day 11-35 after surgery
  Interventions: Drug: Prevention of Venous Thromboembolism; Drug: Placebo Oral Tablet
- Standard of care (Active Comparator): Rivaroxaban from day 3-35 after surgery
  Interventions: Drug: Prevention of Venous Thromboembolism

INTERVENTIONS:
Drug: Prevention of Venous Thromboembolism — Direct oral anticoagulant
  Other Names: Rivaroxaban; Xarelto; anticoag; Direct oral anticoagulant; DOAC
Drug: Placebo Oral Tablet — Placebo
  Arms: Abbreviated lenght of thromboprophylaxis

SUMMARY:
Surgical hip replacement (total hip arthroplasty, THA) is associated with a high risk of venous thromboembolism, but the appropriate duration of postoperative medical thromboprophylaxis ("anticoagulation") remains highly controversial. The international randomized controlled trial (RCT) "ENhanced recovery and ABbreviated LEngth of Anticoagulation for Thromboprophylaxis after primary Hip Arthroplasty" (ENABLE-Hip) will enroll patients undergoing elective THA that are eligible for early mobilization after surgery. The trial will compare a regimen of short-duration (10-day) postoperative anticoagulation (experimental group) to standard-duration (35-day) postoperative anticoagulation (control group) using the direct oral anticoagulant Rivaroxaban (brand name: Xarelto) at the recommended dose. Thus, ENABLE-Hip will be the first major RCT to directly test an overall reduction in the duration of post-THA thromboprophylaxis instead of replacing one antithrombotic drug or regimen by another. Follow-up visits after hospital discharge will be on day 35 and on day 90 after surgery. The primary outcome is acute symptomatic proximal deep vein thrombosis, or symptomatic or fatal pulmonary embolism, within 90 days after surgery. If ENABLE-Hip will demonstrate 'non-inferiority' of the experimental intervention, its benefits will be obvious, as patients are spared many days of unnecessary (and potentially harmful in terms of bleeding risk) anticoagulation.

DETAILED DESCRIPTION:
An increasing proportion of the ageing population in Europe and other parts of the world suffers from hip osteoarthritis and will need surgical joint arthroplasty at some time in their lives. Surgical total hip arthroplasty (THA) is associated with a high risk of venous thromboembolism (VTE), but the appropriate duration of postoperative anticoagulation remains highly controversial. Although current German guidelines continue to advocate anticoagulation for 28-35 days after THA, clinical practice recommendations in other countries are shifting towards much earlier discontinuation of anticoagulants - despite the absence of solid evidence backed by controlled data. The "Enhanced recovery and Abbreviated duration of Anticoagulation for thromboprophylaxis after primary hip Arthroplasty" (ENABLE-Hip) study is a multicentre investigator-initiated and academically sponsored prospective randomised active-control non-inferiority trial. A regimen of short-duration (10-day) prophylactic anticoagulation (experimental arm) will be compared to standard-duration (35-day) anticoagulation as per current guidelines (control arm). Patients will be mobilised early after surgery, following a standardised enhanced recovery protocol. Following randomisation and an initial two-day open-label period of prophylactic anticoagulation as per local protocol, treatment with the study drug (rivaroxaban at the standard, approved prophylactic dose of 10 mg daily) will be started and continued until 10 days after surgery. After this time, patients will be switched (in a double-blinded manner) to placebo in the experimental arm, or continue on active drug in the control arm, until a total of 35 days have elapsed since surgery. The primary outcome is acute symptomatic proximal deep vein thrombosis (DVT), or symptomatic or fatal pulmonary embolism (PE), within the first 3 months after surgery. Participating investigators will be advised to adhere to guideline recommendations regarding clinical suspicion of and diagnostic work-up for VTE. The planned study population of 2,932 patients will provide ≥ 80% power to reject the null hypothesis that δ ≥ 0.01 (where δ = difference between the two arms in symptomatic VTE probability within 3 months) and accept the alternative hypothesis that δ < 0.01, at an overall significance level α = 0.05. A formal interim analysis will be performed after 3-month follow-up of the first 1,760 randomised patients at a significance level α = 0.50, leading to stopping for futility if significance is not obtained, or if recalculation yields an overall sample size of > 3,200 patients. The trial has the potential to inform future national and European guidelines for this large and continuously growing patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age between 18 and 85 years
3. Scheduled to undergo elective unilateral primary THA and eligible for perioperative management based on the ERAS protocol
4. Baseline Timed Up and Go (TUG) test scoring < 20 seconds, corresponding to a good mobility status before surgery
5. Capability to understand and comply with the protocol requirements (e.g., sufficient knowledge of German language to answer the questionnaires, ability to swallow intact capsules).
6. Pregnancy and contraception:

   1. Pregnancy test: Negative serum pregnancy test at screening for women of childbearing potential (WOCBP).
   2. Contraception: WOCBP and men who are able to father a child, willing to be abstinent or use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly beginning at informed consent, for the duration of drug treatment and allowing for a safe wash out period of at least 5 days for female or for male subjects after the last dose of trial medication. This is a very conservative estimate, considering the 'worst case scenario' of a substantially prolonged half-life up to 13 hours (e.g., in older patients and/or those with renal dysfunction) (28), and calculating for at least 8 half-lives to ensure practically non-detectable levels and effects of rivaroxaban.

Exclusion Criteria:

1. Previous DVT or PE
2. Hip or lower limb fracture in the previous three months
3. Major surgical procedure within the previous three months
4. Active cancer defined as metastatic cancer, or cancer requiring chemotherapy or radiation therapy
5. Active peptic ulcer disease, gastritis, or prior gastrointestinal bleeding
6. Obesity with body mass index (BMI) > 40 kg/m2 body surface area
7. Severe renal impairment defined as estimated glomerular filtration rate < 30ml/min
8. Severe hepatic impairment defined as Child Pugh Class B or C
9. Uncontrolled intercurrent illness (i.e., active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, interstitial lung disease, serious gastrointestinal conditions [e.g., diarrhea, malabsorption], psychiatric illness)
10. Active or recent major bleeding at any site, or presence of any major risk factor for bleeding, which, in the judgment of the investigator, may significantly increase the bleeding risk during postoperative anticoagulation treatment
11. Any other medical condition representing a contraindication to discharge within 6 days after surgery
12. Expected requirement for major surgery within a 90-day period post THA
13. Need for long-term anticoagulation (e.g., atrial fibrillation, previous VTE)
14. Need for chronic antiplatelet therapy except for acetylsalicylic acid (ASA) at a dose ≤ 100 mg daily or clopidogrel 75 mg daily
15. Previous participation in this trial
16. Life expectancy < 6 months
17. Participation in another interventional clinical trial within the last 30 days prior to inclusion, unless during the observational follow-up period
18. History of hypersensitivity to the investigational medicinal product (IMP) or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the IMP

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2932 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the rate of acute symptomatic or fatal VTE | within 90 days after surgery
  acute symptomatic or fatal VTE, defined as (i) symptomatic DVT of the popliteal or more proximal leg veins (femoral or iliac veins) or inferior vena cava; or (ii) symptomatic (segmental or more proximal) or fatal PE, occurring in the first 90 days after surgery and confirmed by objective testing.

SECONDARY OUTCOMES:
Length of hospital stay | within 90 days after surgery
  duration of inpatient stay
Changes in patient-reported hip joint-specific disability | within 90 days after surgery
  assessment is made following surgery measured by the HOOS-12 score
Rate of clinically relevant non-major bleedings | within 90 days after surgery
  it does not meet the criteria for major bleeding, but results in hospitalization, aspiration of a wound, or a wound hematoma complicated by infection.
Rate of death from any cause | within 90 days after surgery
  rate of death from any cause
Rate of isolated symptomatic distal DVT | within 90 days after surgery
  rate of symptomatic distal DVT
Rate of myocardial infarction (MI) or stroke | within 90 days after surgery
  rate of MI or stroke
Rate of readmission to the hospital | within 90 days after surgery
  rate of readmissions to the hospital
Number and terms of serious adverse events (SAEs) | within 90 days after surgery
  number of SAEs during study duration
Change in patient mobility | within 90 days after surgery
  measured by Range of motion (ROM) and Timed up and Go (TUG) score
Amount of postoperative healthcare resource utilization | within 35 days after surgery
  visits to health care providers and rehospitalization, employment status
Rate of major bleedings | within 90 days after surgery
  fulfils at least one of the following criteria: (i) fatal (ii) bleeding into a critical area or organ (iii) surgical site bleeding that causes hemodynamic instability (iv) non-surgical site bleeding causing a fall in hemoglobin level of ≥ 20 g L-1, or leading to transfusion of ≥ 2 units of whole blood or red blood cells (v) surgical site bleeding that requires a second intervention (open, arthroscopic, endovascular), or hemarthron of sufficient size to delay mobilization or wound healing
Generic quality of life measured by EQ-5D-5L | within 90 days after surgery
  The EQ-5D is not an abbreviation and is the correct term to use in print or verbally.
  EQ-5D-5L consists of 2 parts:
  1. descriptive system consists of 5 dimensions with 5 levels each. A score of 5 at a minimum means best health state; a score of 25 at a maximum means worst health state.
  2. EQ VAS: a scale from 0 (worst health state) to 100 (best health state) is provided.
  This questionnaire is to be completed by the patient for the current day.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros V. Konstantinides, MD, Univ.-Prof., Study Chair — University Medical Center Mainz, Center for Thrombosis and Hemostasis; Philipp Drees, MD, Univ.-Prof., Study Chair — University Medical Center Mainz, Center for Orthopedics and Trauma Surgery
Locations (6):
- Kepler University Medical Center, Orthopedics and Traumatology, Linz, Upper Austria, Austria
- Germany (5):
  - Sana Clinics Sommerfeld, Dpt. for Surgical Orthopaedics, Kremmen, Brandenburg
  - GPR Rüsselsheim Health and Care Center, Rüsselsheim am Main, Hesse
  - University Medical Center Mainz, Center for Orthopedics and Trauma Surgery, Mainz, Rhineland-Palatine
  - University Medical Center Dresden, University Center for Orthopaedics, Trauma & Plastic Surgery, Dresden, Saxony
  - Evangelical Forest Hospital Berlin - Orthopaedics and Trauma Surgery, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta CR, Pocock SJ. Adaptive increase in sample size when interim results are promising: a practical guide with examples. Stat Med. 2011 Dec 10;30(28):3267-84. doi: 10.1002/sim.4102. Epub 2010 Nov 30. PMID 22105690
- [Background] Mohr K, Mildenberger P, Neusius T, Christodoulou KC, Farmakis IT, Kaier K, Barco S, Klok FA, Hobohm L, Keller K, Becker D, Abele C, Bruch L, Ewert R, Schmidtmann I, Wild PS, Rosenkranz S, Konstantinides SV, Binder H, Valerio L; FOCUS Investigators. Estimated annual healthcare costs after acute pulmonary embolism: results from a prospective multicentre cohort study. Eur Heart J Qual Care Clin Outcomes. 2025 May 1;11(3):334-342. doi: 10.1093/ehjqcco/qcae050. PMID 38950900
- [Background] Klein JP, Logan B, Harhoff M, Andersen PK. Analyzing survival curves at a fixed point in time. Stat Med. 2007 Oct 30;26(24):4505-19. doi: 10.1002/sim.2864. PMID 17348080
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Hood BR, Cowen ME, Zheng HT, Hughes RE, Singal B, Hallstrom BR. Association of Aspirin With Prevention of Venous Thromboembolism in Patients After Total Knee Arthroplasty Compared With Other Anticoagulants: A Noninferiority Analysis. JAMA Surg. 2019 Jan 1;154(1):65-72. doi: 10.1001/jamasurg.2018.3858. PMID 30347089
- [Background] Farmakis IT, Kaier K, Hobohm L, Mohr K, Valerio L, Barco S, Konstantinides SV, Binder H. Healthcare resource utilisation and associated costs after low-risk pulmonary embolism: pre-specified analysis of the Home Treatment of Pulmonary Embolism (HoT-PE) study. Clin Res Cardiol. 2025 Feb;114(2):168-176. doi: 10.1007/s00392-023-02355-5. Epub 2024 Jan 3. PMID 38170252
- [Background] Schoene D, Wu SM, Mikolaizak AS, Menant JC, Smith ST, Delbaere K, Lord SR. Discriminative ability and predictive validity of the timed up and go test in identifying older people who fall: systematic review and meta-analysis. J Am Geriatr Soc. 2013 Feb;61(2):202-8. doi: 10.1111/jgs.12106. Epub 2013 Jan 25. PMID 23350947
- [Background] Prather H, Harris-Hayes M, Hunt DM, Steger-May K, Mathew V, Clohisy JC. Reliability and agreement of hip range of motion and provocative physical examination tests in asymptomatic volunteers. PM R. 2010 Oct;2(10):888-95. doi: 10.1016/j.pmrj.2010.05.005. PMID 20970757
- [Background] Gandek B, Roos EM, Franklin PD, Ware JE Jr. A 12-item short form of the Hip disability and Osteoarthritis Outcome Score (HOOS-12): tests of reliability, validity and responsiveness. Osteoarthritis Cartilage. 2019 May;27(5):754-761. doi: 10.1016/j.joca.2018.09.017. Epub 2018 Nov 10. PMID 30419279
- [Background] Nilsdotter AK, Lohmander LS, Klassbo M, Roos EM. Hip disability and osteoarthritis outcome score (HOOS)--validity and responsiveness in total hip replacement. BMC Musculoskelet Disord. 2003 May 30;4:10. doi: 10.1186/1471-2474-4-10. Epub 2003 May 30. PMID 12777182
- [Background] Blasimann A, Dauphinee SW, Staal JB. Translation, cross-cultural adaptation, and psychometric properties of the German version of the hip disability and osteoarthritis outcome score. J Orthop Sports Phys Ther. 2014 Dec;44(12):989-97. doi: 10.2519/jospt.2014.4994. Epub 2014 Nov 13. PMID 25394689
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Halvorsen S, Mehilli J, Cassese S, Hall TS, Abdelhamid M, Barbato E, De Hert S, de Laval I, Geisler T, Hinterbuchner L, Ibanez B, Lenarczyk R, Mansmann UR, McGreavy P, Mueller C, Muneretto C, Niessner A, Potpara TS, Ristic A, Sade LE, Schirmer H, Schupke S, Sillesen H, Skulstad H, Torracca L, Tutarel O, Van Der Meer P, Wojakowski W, Zacharowski K; ESC Scientific Document Group. 2022 ESC Guidelines on cardiovascular assessment and management of patients undergoing non-cardiac surgery. Eur Heart J. 2022 Oct 14;43(39):3826-3924. doi: 10.1093/eurheartj/ehac270. No abstract available. PMID 36017553
- [Background] Steffel J, Collins R, Antz M, Cornu P, Desteghe L, Haeusler KG, Oldgren J, Reinecke H, Roldan-Schilling V, Rowell N, Sinnaeve P, Vanassche T, Potpara T, Camm AJ, Heidbuchel H; External reviewers. 2021 European Heart Rhythm Association Practical Guide on the Use of Non-Vitamin K Antagonist Oral Anticoagulants in Patients with Atrial Fibrillation. Europace. 2021 Oct 9;23(10):1612-1676. doi: 10.1093/europace/euab065. No abstract available. PMID 33895845
- [Background] Kutzner KP, Meyer A, Bausch M, Schneider M, Rehbein P, Drees P, Pfeil J. Outcome of an "Enhanced Recovery" Program in Contemporary Total Hip Arthroplasty in Germany. Z Orthop Unfall. 2020 Apr;158(2):214-220. doi: 10.1055/a-0946-2523. Epub 2019 Sep 16. English, German. PMID 31525792
- [Background] Matharu GS, Kunutsor SK, Judge A, Blom AW, Whitehouse MR. Clinical Effectiveness and Safety of Aspirin for Venous Thromboembolism Prophylaxis After Total Hip and Knee Replacement: A Systematic Review and Meta-analysis of Randomized Clinical Trials. JAMA Intern Med. 2020 Mar 1;180(3):376-384. doi: 10.1001/jamainternmed.2019.6108. PMID 32011647
- [Background] Lalmohamed A, Vestergaard P, Jansen PA, Grove EL, de Boer A, Leufkens HG, van Staa TP, de Vries F. Prolonged outpatient vitamin K antagonist use and risk of venous thromboembolism in patients undergoing total hip or knee replacement. J Thromb Haemost. 2013 Apr;11(4):642-50. doi: 10.1111/jth.12158. PMID 23387806
- [Background] An VV, Phan K, Levy YD, Bruce WJ. Aspirin as Thromboprophylaxis in Hip and Knee Arthroplasty: A Systematic Review and Meta-Analysis. J Arthroplasty. 2016 Nov;31(11):2608-2616. doi: 10.1016/j.arth.2016.04.004. Epub 2016 Apr 13. PMID 27178011
- [Background] Kapoor A, Ellis A, Shaffer N, Gurwitz J, Chandramohan A, Saulino J, Ishak A, Okubanjo T, Michota F, Hylek E, Trikalinos TA. Comparative effectiveness of venous thromboembolism prophylaxis options for the patient undergoing total hip and knee replacement: a network meta-analysis. J Thromb Haemost. 2017 Feb;15(2):284-294. doi: 10.1111/jth.13566. Epub 2017 Jan 19. PMID 28102615
- [Background] Granziera S, Cohen AT. VTE primary prevention, including hospitalised medical and orthopaedic surgical patients. Thromb Haemost. 2015 Jun;113(6):1216-23. doi: 10.1160/TH14-10-0823. Epub 2015 Mar 26. PMID 25809340
- [Background] CRISTAL Study Group; Sidhu VS, Kelly TL, Pratt N, Graves SE, Buchbinder R, Adie S, Cashman K, Ackerman I, Bastiras D, Brighton R, Burns AWR, Chong BH, Clavisi O, Cripps M, Dekkers M, de Steiger R, Dixon M, Ellis A, Griffith EC, Hale D, Hansen A, Harris A, Hau R, Horsley M, James D, Khorshid O, Kuo L, Lewis P, Lieu D, Lorimer M, MacDessi S, McCombe P, McDougall C, Mulford J, Naylor JM, Page RS, Radovanovic J, Solomon M, Sorial R, Summersell P, Tran P, Walter WL, Webb S, Wilson C, Wysocki D, Harris IA. Effect of Aspirin vs Enoxaparin on Symptomatic Venous Thromboembolism in Patients Undergoing Hip or Knee Arthroplasty: The CRISTAL Randomized Trial. JAMA. 2022 Aug 23;328(8):719-727. doi: 10.1001/jama.2022.13416. PMID 35997730
- [Background] Petersen PB, Kehlet H, Jorgensen CC; Lundbeck Foundation Centre for Fast-track Hip and Knee Replacement Collaborative Group. Safety of In-Hospital Only Thromboprophylaxis after Fast-Track Total Hip and Knee Arthroplasty: A Prospective Follow-Up Study in 17,582 Procedures. Thromb Haemost. 2018 Dec;118(12):2152-2161. doi: 10.1055/s-0038-1675641. Epub 2018 Nov 19. PMID 30453352
- [Background] Jorgensen CC, Jacobsen MK, Soeballe K, Hansen TB, Husted H, Kjaersgaard-Andersen P, Hansen LT, Laursen MB, Kehlet H. Thromboprophylaxis only during hospitalisation in fast-track hip and knee arthroplasty, a prospective cohort study. BMJ Open. 2013 Dec 10;3(12):e003965. doi: 10.1136/bmjopen-2013-003965. PMID 24334158
- [Background] Khan SK, Malviya A, Muller SD, Carluke I, Partington PF, Emmerson KP, Reed MR. Reduced short-term complications and mortality following Enhanced Recovery primary hip and knee arthroplasty: results from 6,000 consecutive procedures. Acta Orthop. 2014 Feb;85(1):26-31. doi: 10.3109/17453674.2013.874925. Epub 2013 Dec 20. PMID 24359028
- [Background] The ICM-VTE Hip & Knee Delegates. Recommendations from the ICM-VTE: Hip & Knee. J Bone Joint Surg Am. 2022 Mar 16;104(Suppl 1):180-231. doi: 10.2106/JBJS.21.01529. No abstract available. PMID 35315610
- [Background] Anderson DR, Dunbar M, Murnaghan J, Kahn SR, Gross P, Forsythe M, Pelet S, Fisher W, Belzile E, Dolan S, Crowther M, Bohm E, MacDonald SJ, Gofton W, Kim P, Zukor D, Pleasance S, Andreou P, Doucette S, Theriault C, Abianui A, Carrier M, Kovacs MJ, Rodger MA, Coyle D, Wells PS, Vendittoli PA. Aspirin or Rivaroxaban for VTE Prophylaxis after Hip or Knee Arthroplasty. N Engl J Med. 2018 Feb 22;378(8):699-707. doi: 10.1056/NEJMoa1712746. PMID 29466159
- [Background] Johanson NA, Lachiewicz PF, Lieberman JR, Lotke PA, Parvizi J, Pellegrini V, Stringer TA, Tornetta P 3rd, Haralson RH 3rd, Watters WC 3rd. Prevention of symptomatic pulmonary embolism in patients undergoing total hip or knee arthroplasty. J Am Acad Orthop Surg. 2009 Mar;17(3):183-96. doi: 10.5435/00124635-200903000-00007. PMID 19264711
- [Background] Jacobs JJ, Mont MA, Bozic KJ, Della Valle CJ, Goodman SB, Lewis CG, Yates AC Jr, Boggio LN, Watters WC 3rd, Turkelson CM, Wies JL, Sluka P, Hitchcock K. American Academy of Orthopaedic Surgeons clinical practice guideline on: preventing venous thromboembolic disease in patients undergoing elective hip and knee arthroplasty. J Bone Joint Surg Am. 2012 Apr 18;94(8):746-7. doi: 10.2106/JBJS.9408.ebo746. No abstract available. PMID 22517391
- [Background] Falck-Ytter Y, Francis CW, Johanson NA, Curley C, Dahl OE, Schulman S, Ortel TL, Pauker SG, Colwell CW Jr. Prevention of VTE in orthopedic surgery patients: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e278S-e325S. doi: 10.1378/chest.11-2404. PMID 22315265
- [Background] Anderson DR, Morgano GP, Bennett C, Dentali F, Francis CW, Garcia DA, Kahn SR, Rahman M, Rajasekhar A, Rogers FB, Smythe MA, Tikkinen KAO, Yates AJ, Baldeh T, Balduzzi S, Brozek JL, Ikobaltzeta IE, Johal H, Neumann I, Wiercioch W, Yepes-Nunez JJ, Schunemann HJ, Dahm P. American Society of Hematology 2019 guidelines for management of venous thromboembolism: prevention of venous thromboembolism in surgical hospitalized patients. Blood Adv. 2019 Dec 10;3(23):3898-3944. doi: 10.1182/bloodadvances.2019000975. PMID 31794602
- [Background] Parvizi J, Ceylan HH, Kucukdurmaz F, Merli G, Tuncay I, Beverland D. Venous Thromboembolism Following Hip and Knee Arthroplasty: The Role of Aspirin. J Bone Joint Surg Am. 2017 Jun 7;99(11):961-972. doi: 10.2106/JBJS.16.01253. No abstract available. PMID 28590382
- [Background] Keller K, Hobohm L, Barco S, Schmidtmann I, Munzel T, Engelhardt M, Goldhofer M, Konstantinides SV, Drees P. Venous thromboembolism in patients hospitalized for hip joint replacement surgery. Thromb Res. 2020 Jun;190:1-7. doi: 10.1016/j.thromres.2020.03.019. Epub 2020 Mar 27. PMID 32247912
- [Background] Cafri G, Paxton EW, Chen Y, Cheetham CT, Gould MK, Sluggett J, Bini SA, Khatod M. Comparative Effectiveness and Safety of Drug Prophylaxis for Prevention of Venous Thromboembolism After Total Knee Arthroplasty. J Arthroplasty. 2017 Nov;32(11):3524-3528.e1. doi: 10.1016/j.arth.2017.05.042. Epub 2017 May 31. PMID 28634095
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Schulman S, Angeras U, Bergqvist D, Eriksson B, Lassen MR, Fisher W; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in surgical patients. J Thromb Haemost. 2010 Jan;8(1):202-4. doi: 10.1111/j.1538-7836.2009.03678.x. Epub 2009 Oct 30. PMID 19878532
- [Background] Mazzolai L, Ageno W, Alatri A, Bauersachs R, Becattini C, Brodmann M, Emmerich J, Konstantinides S, Meyer G, Middeldorp S, Monreal M, Righini M, Aboyans V. Second consensus document on diagnosis and management of acute deep vein thrombosis: updated document elaborated by the ESC Working Group on aorta and peripheral vascular diseases and the ESC Working Group on pulmonary circulation and right ventricular function. Eur J Prev Cardiol. 2022 May 27;29(8):1248-1263. doi: 10.1093/eurjpc/zwab088. PMID 34254133
- [Background] Konstantinides SV, Meyer G, Becattini C, Bueno H, Geersing GJ, Harjola VP, Huisman MV, Humbert M, Jennings CS, Jimenez D, Kucher N, Lang IM, Lankeit M, Lorusso R, Mazzolai L, Meneveau N, Ni Ainle F, Prandoni P, Pruszczyk P, Righini M, Torbicki A, Van Belle E, Zamorano JL; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of acute pulmonary embolism developed in collaboration with the European Respiratory Society (ERS). Eur Heart J. 2020 Jan 21;41(4):543-603. doi: 10.1093/eurheartj/ehz405. No abstract available. PMID 31504429
- [Background] Ghosh A, Best AJ, Rudge SJ, Chatterji U. Clinical Effectiveness of Aspirin as Multimodal Thromboprophylaxis in Primary Total Hip and Knee Arthroplasty: A Review of 6078 Cases. J Arthroplasty. 2019 Jul;34(7):1359-1363. doi: 10.1016/j.arth.2019.03.021. Epub 2019 Mar 13. PMID 30982759
- [Background] Brown GA. Venous thromboembolism prophylaxis after major orthopaedic surgery: a pooled analysis of randomized controlled trials. J Arthroplasty. 2009 Sep;24(6 Suppl):77-83. doi: 10.1016/j.arth.2009.06.002. Epub 2009 Jul 22. PMID 19628366
- [Derived] Drees P, Schmidtmann I, Herbst M, Becker D, Barco S, Klok FA, Keller K, Hobohm L, Christodoulou KC, Abele C, Bauersachs R, Ageno W, Grove EL, Kehlet H, Hufen F, Klonschinski T, Afghanyar Y, Eckhard L, Martin N, Fischer S, Gorbulev S, Rath D, Mavromanoli AC, Jabbour C, Lang I, Couturaud F, Heiss C, Binder H, Konstantinides S. Enhanced recovery and abbreviated length of anticoagulation for thromboprophylaxis after primary hip arthroplasty rationale and design of the ENABLE-hip trial. J Thromb Thrombolysis. 2025 Aug;58(6):689-698. doi: 10.1007/s11239-025-03110-5. Epub 2025 May 29. PMID 40442449